CLINICAL TRIAL: NCT05202457
Title: Review of Outcomes in Patients With Cirrhosis Undergoing General Surgery
Brief Title: Cirrhotics Undergoing General Surgery
Status: Completed | Type: Observational
Sponsor: Danny Lascano (Other)
Responsible Party: Sponsor-Investigator, Danny Lascano, Research Resident, Westchester Medical Center
Organization: Westchester Medical Center (Other)
Other Study IDs: L12-124
Record Dates: First submitted 2022-01-05; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Cirrhosis, Liver
Keywords: elective surgery; cirrhotics; cirrhosis
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis | interventions — Elective Surgical Procedures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cirrhosis: Patients with cirrhosis undergoing urgent and elective surgery
  Interventions: Procedure: Elective surgery

INTERVENTIONS:
Procedure: Elective surgery — Patient undergoing elective or urgent surgery

SUMMARY:
Surgery on cirrhotic patients represents a clinical challenge but intervening before these patients develop complications can prolong the likelihood of these patients making it to transplant for those transplant-eligible candidates. There is no literature on survival to transplant afforded by surgery nor 90 day and 1-year outcomes after any surgical procedures on this population. The investigator's aim is to study the principal investigator's single surgical center experience at a tertiary hospital with the largest referral center in the area for liver transplant candidates. The investigators hypothesize, that although the risk is high for patients undergoing surgery it is much lower than historically reported, may make more patients eligible for transplant and prevent complications that may lead to death for the transplant eligible, and may reveal associations that can lead to good outcomes in this high-risk population.

DETAILED DESCRIPTION:
Introduction

The incidence of cirrhosis is increasing as alcoholic liver disease overtakes hepatitis as the cause of cirrhosis although it will likely stabilize as Hepatitis C treatment makes its way through the population. However, liver disease continues to have a large impact on morbidity and mortality with a prevalence of approximately 4.5 million people diagnosed with liver disease with an incidence of 1.8% per year and 12.8 deaths per 100,000 people. The cost of treating cirrhosis ranges from $14 million to $2 billion dollars depending on the etiology of the disease. The large cost is driven by multiple hospitalizations, surgical procedures, rehabilitation/nursing home, and other factors.

For surgeons, cirrhotic patients represent an especially high-risk patient population. In the past, many surgeons were hesitant to offer definitive surgeries for symptomatic cholelithiasis, hernias, or cancer surgeries. Historically these patients had a high risk of mortality with competing causes of mortality driven by liver cirrhosis as well as other issues. Hence, it was thought that these patients should only be operated on in emergent cases unless it precluded them from being transplant eligible. For example, Garrison, et al. noted in 1984 that patients who underwent exploratory laparotomy with either a Child B and C had a 31% and 76% mortality, respectively. Furthermore, this was not unique to that group as another group in 1997 showed surgeries like hernia procedures, cholecystectomy, and other procedures had mortality rates of up to 82% for Child C cirrhotics. As general post-surgical care and critical care have improved, contemporary studies show that mortality although decreased still is significant. A prospective study looking at cirrhotic patients who underwent an umbilical hernia for 30 patients had a mortality of 6%. Moreover, a retrospective analysis of a prospectively maintained database from the American College of Surgeons National Surgical Quality Improvement Program revealed that in a series of 390 pts undergoing umbilical hernia repair there was a 5.1% mortality and 13.1% morbidity in comparison to 0.1 and 3.9% on non-cirrhotic patients, respectively.

There are few papers that look at the drivers of morbidity, mortality, and complications among this population and none looking at more than 30 days post-operative re-admissions, morbidity, or mortality. Furthermore, there is no literature on how elective or emergent surgery may facilitate a longer survival so that patients may still be alive and eligible to receive their liver, the ultimate treatment for liver cirrhosis. Hence, the investigator's tertiary center experience was evaluated focusing on pre-operative, intraoperative, and postoperative factors that may explain the drivers of morbidity and mortality in cirrhotics undergoing elective and emergent surgery. The investigators will also study at how many patients after their index procedure survived to receive their liver transplant. Hence, the investigator's surgical, single-center experience at a tertiary hospital with the largest referral center in the area for liver transplant candidates for any cirrhotics requiring surgery either emergent (<24 hours since admission), urgent (same admission but > 24 hrs), or elective (patient coming from outpatient setting for planned surgery). The investigators hypothesize, that although the risk is high for patients undergoing surgery, it currently is much lower than historically reported, which may make more patients eligible for transplant and prevent complications that may lead to death for the transplant eligible patients, and may reveal associations that can lead to good outcomes in this high-risk population.

Materials and Methods

The investigator's institutional review board approved this study and data were collected in a retrospective fashion. Initially, a query was done looking at all participants with cirrhosis who underwent any procedure done by the principal investigator. After this, a chart review was done looking at all the participants with a diagnosis of cirrhosis via manual chart review. The index procedure, as well as any re-operation done, were included and all performed by the surgeon who is the principal investigator. Furthermore, pre-operative data that was collected included medications used to treat cirrhosis, etiology of cirrhosis, biological Na-MELD/ Child's classification, whether a transjugular intrahepatic portosystemic shunt was performed, the incidence of esophageal varices/ ascites, pre-operative drainage of ascites or placement of a drain as well as cases of refractory ascites.

Furthermore, intraoperative data were obtained from the anesthesia records regarding estimated blood loss, crystalloid/ colloid administered, blood products administered, any episodes of hypotension, and the use of vasopressors. Post-operative data collected included any complications, blood products administered, the use of colloids, and finally the date of discharge. The participants were tracked for over a year and any cases of re-admission were noted from the charts and the causes of re-admission were noted for further analysis.

Data was collected in a de-identified fashion. Comparisons were done via Student T-tests when applicable. Logistic regression was done to identify factors associated with a given outcome including morbidity and mortality with a limit of 3 factors chosen in a univariable model and multivariable model given the low number of cases. Kaplan Meier curves were done to analyze the time to transplant after elective surgery to analyze whether elective surgery may increase the life span of cirrhotics who undergo surgery and stratifying by different risk factors to predict who may need a transplant sooner after elective surgery. Data were analyzed via SPSS 26.0.

ELIGIBILITY:
Inclusion Criteria:

* All non-transplant surgical procedures by the principal investigator over a 5-year period (2013-2018)
* Patients with a known, symptomatic and documented pre-operative history of cirrhosis

Exclusion Criteria:

* Asymptomatic or incidentally discovered cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years or over who presented to Westchester Medical Center, a quaternary hospital system in the Hudson Valley
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Number of patients that die at 30, 90 and 365 days after index surgery | 1 year
  Death within 30, 90 and 365 days after surgery

SECONDARY OUTCOMES:
Number of patients that have a complication at 30, 90 and 365 days after index surgery | 1 year
  Complications within 30, 90 and 365 days after surgery
Number of patients that receive a liver transplant after their index surgery | 1 year
  Number of patients who make it to surgery af their index surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Veillette, MD, Principal Investigator — Westchester Medical Center
Locations (1):
- Westchester Medical Center, Valhalla, New York, United States

IPD SHARING:
Plan to Share IPD: No
Given the low number of patients and risk of identification, decision has been made not to share this data.

REFERENCES:
- [Background] Neff GW, Duncan CW, Schiff ER. The current economic burden of cirrhosis. Gastroenterol Hepatol (N Y). 2011 Oct;7(10):661-71. PMID 22298959
- [Background] Garrison RN, Cryer HM, Howard DA, Polk HC Jr. Clarification of risk factors for abdominal operations in patients with hepatic cirrhosis. Ann Surg. 1984 Jun;199(6):648-55. doi: 10.1097/00000658-198406000-00003. PMID 6732310
- [Background] Mansour A, Watson W, Shayani V, Pickleman J. Abdominal operations in patients with cirrhosis: still a major surgical challenge. Surgery. 1997 Oct;122(4):730-5; discussion 735-6. doi: 10.1016/s0039-6060(97)90080-5. PMID 9347849
- [Background] Eker HH, van Ramshorst GH, de Goede B, Tilanus HW, Metselaar HJ, de Man RA, Lange JF, Kazemier G. A prospective study on elective umbilical hernia repair in patients with liver cirrhosis and ascites. Surgery. 2011 Sep;150(3):542-6. doi: 10.1016/j.surg.2011.02.026. Epub 2011 May 31. PMID 21621237
- [Background] Cho SW, Bhayani N, Newell P, Cassera MA, Hammill CW, Wolf RF, Hansen PD. Umbilical hernia repair in patients with signs of portal hypertension: surgical outcome and predictors of mortality. Arch Surg. 2012 Sep;147(9):864-9. doi: 10.1001/archsurg.2012.1663. PMID 22987183
- See also: Data regarding incidence/ prevalence of cirrhosis in the US — https://ftp.cdc.gov/pub/Health_Statistics/NCHS/NHIS/SHS/2018_SHS_Table_A-4.pdf
- See also: Kochanek K.K. MSL, Xu J., Arias E. Deaths: Final Data for 2017. National Vital Statistics Reports, [Internet]. 2017; 68(9):[77 p.]. Available from: https://http://www.cdc.gov/nchs/data/nvsr/nvsr68/nvsr68_09-508.pdf — http://www.cdc.gov/nchs/data/nvsr/nvsr68/nvsr68_09-508.pdf